CLINICAL TRIAL: NCT03785626
Title: Quantitative Prediction of Carotid Endarterectomy Risk Based on Vascular Structure and Hemodynamics by Vascular Ultrasound Evaluation System
Brief Title: Risk Prediction of Carotid Endarterectomy by Vascular Ultrasound Evaluation
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: VUS-CEA
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Stroke
Keywords: Ultrasound; Carotid Endarterectomy; Risk Prediction Model
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CEA surgery — patients with carotid artery severe (70-99%) stenosis or occlusion received CEA surgery

SUMMARY:
Carotid endarterectomy (CEA) is one of the surgical treatment methods for the reconstruction of arterial stenosis or occlusion. Perioperative stroke, cerebral hemorrhage,hyperperfusion syndrome and death are main complications of CEA. Investigator have established a risk prediction model of the procedure based on vascular characteristics and hemodynamic parameters retrospectively. This prospective study was aimed to verify the predictive ability of CEA comprehensive prediction model through the analysis of patients receiving CEA procedure in the investigator's center in the next two years.

DETAILED DESCRIPTION:
Subjects: In this study, a total of 600-800 patients with severe carotid artery stenosis or occlusion who scheduled for CEA are recruited.

Data collection:

1. The plaque characteristics, stenosis degrees of carotid artery and intracranial arteries, and collateral circulation are evaluated by ultrasound prior to the procedure.
2. CT, MRI and digital subtraction angiography (DSA) were applied pre- and post-procedure to identify the clinical events.

Endpoint: The combination endpoints events of death, cerebral hemorrhage , newly cerebral infarction, hyperperfusion syndrome within 30-day after the procedure.

Statistical analysis plans: The Statistical Package of Social Sciences (SPSS version 22.0) software are used for statistical analysis. The area under the receiver operating characteristic (ROC) curve and hosmer-lemeshow test were used to evaluate the discrimination and calibration of the risk prediction model.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with carotid artery severe (70-99%) stenosis or occlusion diagnosed by color duplex flow imaging (CDFI) and confirmed by CT angiography (CTA) or digital subtraction angiography (DSA).
2. Patient has the indications for carotid artery stenting or CEA according to the guidelines published by the Stroke Prevention Engineering Committee, the National Health Commission of China.
3. MRI and CT were applicated pre- and postoperation.

Exclusion Criteria:

1. Patients with non-atherosclerotic carotid artery stenosis or occlusion, such as dissection, aneurysm, arteritis, cardiac embolism, et al.
2. Lack of any imaging evaluation results, such as ultrasound, MRI or CT.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carotid artery severe (70-99%) stenosis or occlusion who are scheduled for CEA.
Sampling Method: Non-Probability Sample
Enrollment: 1498 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The rate of death, stroke or hemorrhage | 30 days postoperation
  The rate of combination endpoints events of death, cerebral hemorrhage , newly cerebral infarction, hyperperfusion syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No